CLINICAL TRIAL: NCT03604120
Title: PREOPTI-DAM: High-flow Nasal Cannula Oxygen Versus Standard Oxygenation During Intubation for Patient at Risk of Difficult Intubation: A Randomized Controlled Clinical Trial
Brief Title: Preoxygenation for Difficult Airway Management
Acronym: PREOPTI-DAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC17_0474
Record Dates: First submitted 2018-06-22; First posted 2018-07-27 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Intubation;Difficult
Keywords: Preoxygenation; High flow nasal cannula

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preoxygenation with high flow therapy by nasal cannula (Experimental): High flow oxygen therapy by nasal cannula.
  Interventions: Device: Preoxygenation with high flow therapy by nasal cannula
- Preoxygenation by standard Facial mask (Active Comparator): Patients randomized in "STANDARD FACIAL MASK" group will receive a four minutes preoxygenation period with a standard face mask (15 l/mn) before orotracheal intubation under laryngoscopy after crash induction or Fiber-optic intubation under spontaneous ventilation.
  Interventions: Device: Preoxygenation by standard Facial mask

INTERVENTIONS:
Device: Preoxygenation with high flow therapy by nasal cannula — Preoxygenation during 4 minutes with High Flow Nasal Cannula (60l/min FiO2 = 1) before fiber-optic or laryngoscopic intubation. The device will be maintained in place throughout the intubation procedure in order to achieve oxygenation.
  Arms: Preoxygenation with high flow therapy by nasal cannula
Device: Preoxygenation by standard Facial mask — * For Fiber-optic intubation: patients will receive a 4 minutes FIBROXY facial mask preoxygenation with FiO2=100%. The FIBROXY facial mask will be maintained in place during the intubation procedure.
  * For Laryngoscopic intubation: patients will receive a 4 minutes standard facial mask preoxygenation with FiO2=100%. The standard facial mask will be removed after crash induction to proceed to intubation.
  Arms: Preoxygenation by standard Facial mask

SUMMARY:
Tracheal intubation in operating room for patients at risk of difficult intubation remains a critical event. The aim of this study is to determine whether Nasal High Flow Therapy by nasal cannula Optiflow® administered before and during intubation is more efficient than the standard care for pre-oxygenation and oxygenation during anticipated difficult intubation

DETAILED DESCRIPTION:
This study will be designed as followed: Patients will be randomized in 2 groups:

* Preoxygenation during 4 minutes with High Flow Nasal Cannula (60l/min FiO2 = 1) before and during intubation. The device will be maintained in place throughout the intubation procedure (including fiber-optic or laryngoscopic) in order to achieve oxygenation.
* Or Standard Preoxygenation during 4 minutes with FIBROXY® (Fiber-optic intubation) or standard facial mask (Laryngoscopic intubation), at FiO2=100%. FIBROXY mask will be maintained in place during the fiberoptic procedure. Standard facial mask, will be removed after the crash induction.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of aged and over
* And anticipated difficult intubation
* And requiring a rapid sequence induction for laryngoscopic intubation
* Or requiring a fiberoptic intubation

Exclusion Criteria:

* BMI > 35
* Pulse oxymetry < 90% in ambient air
* Haemodynamic instability
* Pregnancy
* Protected adult
* Lack of consent
* Patient already enrolled in another randomized study looking forward improving preoxygenation quality.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2018-09-19 (Actual); Primary Completion 2021-03-08 (Actual); Study Completion 2021-03-08 (Actual)

PRIMARY OUTCOMES:
Incidence of desaturation below 95% or manual facial mask reventilation during ETI procedure. | 4 minutes
  To determine whether High-Flow nasal cannula used for preoxygenation and oxygenation during intubation, is more efficient than standard care during difficult intubation. This outcome will be assessed from the beginning of the preoxygenation period to the end of orotracheal intubation by monitoring the pulse oxymetry.

SECONDARY OUTCOMES:
Improvement of quality of preoxygenation | 4 minutes
  duration of proceedings
Reduction in side effects incidence related to intubation | 6 hours
Morbi-mortality during surgery. | 6 hours
  Per and postoperative complication rate

CONTACTS AND LOCATIONS:
Overall Officials: Mickael VOURC'H, PH, Principal Investigator — Nantes University Hospital
Locations (1):
- Nantes University Hospital, Nantes, France

REFERENCES:
- [Derived] Vourc'h M, Huard D, Le Penndu M, Deransy R, Surbled M, Malidin M, Mahe PJ, Guitton C, Roquilly A, Malard O, Feuillet F, Rozec B, Asehnoune K. High-flow oxygen therapy versus facemask preoxygenation in anticipated difficult airway management (PREOPTI-DAM): an open-label, single-centre, randomised controlled phase 3 trial. EClinicalMedicine. 2023 May 22;60:101998. doi: 10.1016/j.eclinm.2023.101998. eCollection 2023 Jun. PMID 37251624
- [Derived] Vourc'h M, Huard D, Feuillet F, Baud G, Guichoux A, Surbled M, Tissot M, Chiffoleau A, Guitton C, Jaber S, Asehnoune K. Preoxygenation in difficult airway management: high-flow oxygenation by nasal cannula versus face mask (the PREOPTIDAM study). Protocol for a single-centre randomised study. BMJ Open. 2019 Apr 25;9(4):e025909. doi: 10.1136/bmjopen-2018-025909. PMID 31028041